CLINICAL TRIAL: NCT06120478
Title: The Second Affiliated Hospital of Air Force Military Medical University
Brief Title: Prediction of Risk Factors for Adverse Events After Head and Neck Vascular Recanalization Surgery Based on Machine Learning Models
Status: Completed | Type: Observational
Sponsor: Tang-Du Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Bei Liu
Record Dates: First submitted 2023-11-02; First posted 2023-11-07 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Machine Learning

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- xi'an
  Interventions: Other: observe
- shanxi
  Interventions: Other: observe

INTERVENTIONS:
Other: observe — observational study

SUMMARY:
Prediction of risk factors for adverse events after head and neck vascular recanalization surgery based on machine learning models

ELIGIBILITY:
Inclusion Criteria:

* All enrolled patients were diagnosed with clear head and neck artery stenosis and a risk event after head and neck revascularization;
* Location of lesion: origin of internal carotid artery, bifurcation of internal and external carotid arteries;
* Patients with symptomatic head and neck artery stenosis and dangerous events after head and neck blood flow reconstruction, and with a degree of stenosis ≥ 70% on non-invasive examination or stenosis ≥ 50% found on angiography;
* Asymptomatic head and neck artery stenosis and risk events after head and neck revascularization, with a degree of stenosis ≥ 70% on non-invasive examination or stenosis ≥ 60% found on angiography;
* Asymptomatic head and neck artery stenosis and dangerous events after head and neck blood flow reconstruction, with a non-invasive examination of stenosis degree less than 70%, but angiography or other examinations indicate that the stenosis lesion is in an unstable state;
* Symptomatic head and neck artery stenosis and risk events after head and neck revascularization, non-invasive examination of head and neck artery stenosis and risk events after head and neck revascularization are 50% to 69%;
* Sign the project informed consent form

Exclusion Criteria:

* Patients with poor overall condition and intolerance to general anesthesia;
* Patients with mental illness or severe mental illness;
* Severe respiratory system diseases;
* Pregnant and lactating women;
* Participating in another clinical study;
* Patients with advanced tumors or those who are expected to die within one year;

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing vascular recanalization surgery due to stroke
Sampling Method: Non-Probability Sample
Enrollment: 1300 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
death | one year

SECONDARY OUTCOMES:
Recurrence of stroke | one year

CONTACTS AND LOCATIONS:
Locations (1):
- Tangdu Hospital, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Yes